CLINICAL TRIAL: NCT04308408
Title: Front of Pack Nutritional Labeling of Processed Foods Among Mexican Consumers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, Alejandra Jáuregui de la Mota, Chair of the Department of Physical Activity and Healthy Lifestyles, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 7-68S4-17
Record Dates: First submitted 2020-03-10; First posted 2020-03-16 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Food Labeling
Keywords: food labeling; nutritional quality; label understanding; purchasing behavior
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mexican Guideline Daily Allowance (GDA) (Active Comparator): Guideline Daily Amounts (GDA) is a purely numerical and reductive labeling system, indicates the grams and percentages (according to the guideline-based daily intakes) per portion of kilocalories, saturated fats, other fats, sugars, and sodium, with no specific judgement, opinion or recommendation.
  Interventions: Behavioral: Guideline Daily Amounts; Behavioral: Video
- Ecuador's Multiple Traffic Light (MTL) (Experimental): Multiple traffic light labels, an interpretive nutrient-specific FOP label, use the typical traffic light colors (green, yellow/amber, red) and text descriptors to indicate the high, medium, or low content of total fat, sugar and salt.
  Interventions: Behavioral: Multiple Traffic Light; Behavioral: Video
- Chilean Warning Labels in Red (Experimental): Warning Labels (WL), another nutrient-specific interpretive FOP labelling scheme, include 'high in' symbols for products that exceed limits of energy, sodium, sugar and saturated fat.
  Interventions: Behavioral: Warning Labels; Behavioral: Video

INTERVENTIONS:
Behavioral: Guideline Daily Amounts — All food items displayed the corresponding GDA label in the lower left corner of the front of the package.
  Arms: Mexican Guideline Daily Allowance (GDA)
Behavioral: Multiple Traffic Light — All food items displayed the corresponding MTL label in the lower left corner of the front of the package.
  Arms: Ecuador's Multiple Traffic Light (MTL)
Behavioral: Warning Labels — Food products were labeled with "High in" labels In the lower left corner of the front of the package. In total, 37 of the 60 food products in the shopping site did not display a WL.
  Arms: Chilean Warning Labels in Red
Behavioral: Video — Participants viewed a short (less than 1 min) video explaining how to interpret the label.

SUMMARY:
The effect of three front of pack (FOP) labeling schemes (Mexican Guideline Daily Amounts (GDA), Ecuador's Multiple Traffic Light (MTL) and Chilean Warning Labels (WL) in red) on purchasing intentions was evaluated using a randomized experiment of an online shopping simulation. The study employed an online grocery store developed for this purpose to simulate a shopping situation.

DETAILED DESCRIPTION:
Nutrition labels may modify purchasing behavior. Different labels may influence consumer purchasing behaviors in different ways.

In general, for nutrition labels to have any effect on purchasing decisions, consumers must first be exposed to them and perceive the displayed information on the labels. Then, the effect will be mediated by consumer understanding. Based on this understanding, consumers may use the label to make inferences about the nutritional quality or healthiness of the product, which, together with other information (e.g. trust or liking of the label or taste of the product) may affect the evaluation of the product and eventually the purchase decision of the product.

GDA provide numeric information on the content of key nutrients in the food product without interpreting the information.

MTL and WL are nutrient-specific labels providing an interpretation of the nutritional content of specific nutrients in the product. The MTL uses traffic light colors to indicate the high (red) or low (green) content of key nutrients, whereas the WL are only included in a product when the content of each key ingredient is above specific criteria.

Trained undergraduate student research assistants from eight universities across the country recruited the study participants. Research assistants were trained on how to approach and recruit participants and obtain informed consent. They were instructed to recruit 20 or more participants each. Recruitment took place in public spaces previously selected by convenience by the research team, based on their use by low- and middle-income groups in Mexico (i.e., public schools, public squares, public health centers, as well as supermarket chains and shopping centers located in low-income neighborhoods). Potential participants were approached by research assistants, who explained study objectives and invited them to be part of the study. Then, individuals were screened for eligibility using a 3-item screener. To access this screener, research assistants used a tablet or laptop with internet-access, to access a unique web address where our web-based tool was hosted. Research assistants were automatically informed by the web-based tool about the eligibility of the participant. Informed consent was obtained from all eligible participants using an automated computer-based form. Then, the tablet or laptop was handed to participants, who completed a self-administered online demographic and health survey, and then accessed the online shopping site to simulate a shopping situation. Participants completed the shopping task on the same day at the public place where they were recruited.

After allocation, participants viewed a video explaining how to correctly interpret the assigned label. Each participant was asked to shop freely, to better mimic real-world grocery shopping conditions. Research assistants instructed participants as follows: "take into account the assigned label and choose your preferred products". Participants were assigned an initial budget to do their shopping, although they did not pay actual money for their groceries. This budget corresponded to their weekly expenditure in groceries reported in the demographic survey, from 500-5000 Mexican pesos ($28-280 USD), in multiples of 500. No specific instructions were given related to the number or total cost of food products purchased.

FOP nutrition labels were affixed on the food items of the virtual supermarket. The store displayed the name, price and the front of the pack image of 60 food products from 5 food groups (ready-made foods, dairy products, non-dairy beverages, salty snacks, and breakfast cereals). Products were shown on traditional shopping shelves. Participants could zoom in to look more closely at the products and their prices, and could click on the product to access a new pop-up window. This new window displayed product information (i.e., name and brand), a larger image of the front of the product packaging, and an area where they could select the amount or number of products they wanted to put in their shopping cart. The pop-up window was the only way in which participants could select the food products to "purchase". Participants could also zoom in further on this pop-up to look more closely at the package and the nutritional label.

After completing their shopping, participants revised their shopping cart and "purchased" their products. A brief feedback on the nutritional quality of the products in their shopping cart was provided as a retribution for their time.

ELIGIBILITY:
Inclusion Criteria:

* Consuming at least one of the five food groups included in the shopping site (salty snacks, beverages, dairy products, breakfast cereals and ready-made foods)
* Shopping for groceries at least twice per week

Exclusion Criteria:

* Working in the food and beverage industry
* Having any of their direct family members working in the food and beverage industry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2105 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Mean nutritional quality of the shopping cart | On the date of randomization
  The Nutrient Profiling Scoring Criterion model was used as the main measure to evaluate the nutritional quality of the shopping cart.
Mean nutritional quality of the shopping cart (negative nutrients) | On the date of randomization
  The Nutrient Profiling Scoring Criterion baseline score, considering only negative nutrients, was used to explore a nutritional quality measure consistent with the key nutrients evaluated.

SECONDARY OUTCOMES:
Mean protein content | On the date of randomization, after completion of the online shopping simulation
  The mean protein content per 100g or 100 mL of the purchased items was calculated by dividing the total protein content in the shopping cart by the number of products purchased
Mean fiber content | On the date of randomization, after completion of the online shopping simulation
  The mean fiber content per 100g or 100 mL of the purchased items was calculated by dividing the total fiber content in the shopping cart by the number of products purchased
Mean sodium content | On the date of randomization, after completion of the online shopping simulation
  The mean sodium content per 100g or 100 mL of the purchased items was calculated by dividing the total sodium content in the shopping cart by the number of products purchased
Mean sugar content | On the date of randomization, after completion of the online shopping simulation
  The mean sugar content per 100g or 100 mL of the purchased items was calculated by dividing the total sugar content in the shopping cart by the number of products purchased
Mean saturated fat content | On the date of randomization, after completion of the online shopping simulation
  The mean saturated fat content per 100g or 100 mL of the purchased items was calculated by dividing the total saturated fat content in the shopping cart by the number of products purchased.
Mean energy content | On the date of randomization, after completion of the online shopping simulation
  The mean energy content per 100g or 100 mL of the purchased items was calculated by dividing the total energy content in the shopping cart by the number of products purchased
Mean fat content | On the date of randomization, after completion of the online shopping simulation
  The mean fat content per 100g or 100 mL of the purchased items was calculated by dividing the total fat content in the shopping cart by the number of products purchased
Time to first product selection (minutes) | On the date of randomization, during the online shopping simulation
  Calculated as the time required to "buy" a product after entering the online grocery store.
Time spent looking at a product before deciding to buy it (seconds) | On the date of randomization, during the online shopping simulation
  Estimated as the time between observing the food product on the pop-up window and clicking on the "add to shopping cart" button
Time spent looking at a product before deciding not to buy it (seconds) | On the date of randomization, during the online shopping simulation
  Estimated as the time between observing the food product on the pop-up window and going back to the shopping shelf
Total time spent shopping (minutes) | On the date of randomization, after completion of the online shopping simulation
  Calculated as the time spent shopping, between entering and exiting the online grocery store.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Jauregui, ScD, Principal Investigator — Instituto Nacional de Salud Pública
Locations (8):
- Mexico (8):
  - Hospital de Alta Especialidad del Bajío, León, Guanajuato
  - Universidad Autónoma Metropolitana, Mexico City, Mexico City
  - Univesidad Autónoma de Morelos, Cuernavaca, Morelos
  - Universidad Autónoma de Nuevo León, Monterrey, Nuevo León
  - Universidad de Monterrey, Monterrey, Nuevo León
  - Universidad Iberoamericana, Mexico City
  - Universidad Nacional Autónoma de México, Mexico City
  - Universidad Autónoma de San Luis Potosí, San Luis Potosí City

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years after completion of recruitment
Access Criteria: Data access requests will be reviewed by the principal investigator. Requestors will be required to sign a Data Acess agreement.

REFERENCES:
- [Derived] Jauregui A, Vargas-Meza J, Nieto C, Contreras-Manzano A, Alejandro NZ, Tolentino-Mayo L, Hall MG, Barquera S. Impact of front-of-pack nutrition labels on consumer purchasing intentions: a randomized experiment in low- and middle-income Mexican adults. BMC Public Health. 2020 Apr 6;20(1):463. doi: 10.1186/s12889-020-08549-0. PMID 32252716

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT04308408/Prot_SAP_000.pdf